CLINICAL TRIAL: NCT03210233
Title: Development of a Novel Diagnostic Pathway for Immediate Type Hypersensitivity Reactions to Teicoplanin, Including Invivo and Ex-vivo Testing Modalities.
Brief Title: Development of Diagnostic Pathway for Teicoplanin Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AN15/424
Record Dates: First submitted 2017-03-27; First posted 2017-07-06 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Hematologic Tests; Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Naive controls (Experimental): Never received teicoplanin. Blood test, skin testing and challenge testing.
  Interventions: Procedure: Blood test, skin testing and challenge testing.
- High Risk (Experimental): Received teicoplanin and suffered suspected IgE mediated anaphylaxis. Blood test, skin testing and challenge testing.
  Interventions: Procedure: Blood test, skin testing and challenge testing.
- Low Risk (Experimental): Received teicoplanin previously with no adverse reaction Blood test, skin testing and challenge testing.
  Interventions: Procedure: Blood test, skin testing and challenge testing.

INTERVENTIONS:
Procedure: Blood test, skin testing and challenge testing. — Skin Prick Testing (SPT) and Intradermal Testing (IDT). We will follow the STARD framework for reporting studies of diagnostic accuracy

SUMMARY:
Teicoplanin is an antibiotic used very commonly to prevent infection during surgery. Its use has expanded rapidly in the last few years, with around 18,500 doses administered in Leeds Teaching Hospitals NHS Trust alone, in 2014-15. Unfortunately, anaphylaxis (a severe allergic reaction) to the drug appears to be increasing. These reactions can result in admission to intensive care, prolong hospital stay, or even be fatal.

It is vital that patients who suffer anaphylaxis have tests to accurately identify the cause, so they can avoid the drug in future. However these tests are currently very limited, because we don't have any diagnostic tools proven to confirm or refute a diagnosis of teicoplanin allergy. We have to make a 'best guess' diagnosis, leaving patients vulnerable to harm in the future, should they require antibiotics again. We need to reliably diagnose teicoplanin allergy to reduce this arm. Where a diagnosis of teicoplanin allergy is confirmed, patients and their doctors know to avoid it. Importantly, where allergy is excluded, teicoplanin can be safely used, avoiding alternatives that may be less effective, more toxic, and more expensive. This directly benefits individuals, saves the NHS money by reducing avoidable harm, and helps improve antibiotic stewardship at a population level - which in the long term helps reduce antibiotic resistance. The clinical need for this work has become imperative.

Collaborating with our industry partner ThermoFisher (significant expertise in this area), we aim to:

1. Standardise the current skin testing protocols being used when testing patients with suspected teicoplanin allergy.
2. Develop laboratory tests to support the skin tests, and give a more confident diagnosis to patients.
3. Understand how and why people develop allergy to teicoplanin, to better predict and modify the allergic response.

ELIGIBILITY:
Inclusion Criteria:

All groups >16 years, willing and able to give informed consent.

Group 1(G1). Naïve controls 72 recruited from staff/students of the University of Leeds (n= >40,000 persons) where infrastructure exists to advertise and rapidly recruit

INCLUSION CRITERIA:

* >16 years, willing and able to give informed consent
* Never received teicoplanin

Group 2(G2). "High risk". Received teicoplanin and suffered IgE mediated allergic reaction as defined by our pre-set clinical criteria n=132 to achieve n-119 with complete follow up data, recruited from the "Suspected Anaesthetic Allergy clinic", where patients who have suffered suspected perioperative allergy are referred.

INCLUSION CRITERIA:

* >16 years, willing and able to give consent
* Received teicoplanin and suffered suspected IgE mediated anaphylaxis

Group 3 (G3). "Low risk". Received teicoplanin without reaction

G3: n=397 to achieve n=357 with complete follow up data, recruited from surgical areas where teicoplanin is used routinely; predominantly orthopaedic surgery

Exclusion Criteria:

EXCLUSION CRITERIA for G1, G2 and G3.

* History of antibiotic anaphylaxis/specialist drug allergy testing
* History of toxic epidermal necrolysis or Stevens Johnson syndrome
* Brittle asthma
* Dermographism or other poorly controlled skin condition
* Pregnant, planning to become pregnant during study, breastfeeding

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
In vivo testing | 12 months
  Skin testing protocols, which identify IgE mediated sensitivity to teicoplanin.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No